CLINICAL TRIAL: NCT04451941
Title: Determination of Clinical Effects of Brain Machine Interface in Chronic Stroke Patient Without Wrist Extensor Strength
Brief Title: Clinical Effects of Brain Machine Interface in Chronic Stroke Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Chief of Brain Injury Rehabilitation Department, Principal Investigator, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2020-01-007
Record Dates: First submitted 2020-06-04; First posted 2020-06-30 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: brain machine interface; chronic stroke; wrist extensor strength
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RecoveriX with individual EEG calibration (Experimental): RecoveriX applied functional electrical stimulation (FES) according to individual brainwave by individual EEG calibration for 4 weeks
  Interventions: Device: Experimental: RecoveriX with individual EEG calibration
- RecoveriX without individual EEG calibration (Sham Comparator): RecoveriX applied FES according to the brainwave of other subjects regardless of the individual brainwave for 4 weeks
  Interventions: Device: RecoveriX without individual EEG calibration

INTERVENTIONS:
Device: Experimental: RecoveriX with individual EEG calibration — RecoveriX applied FES according to individual brainwave by individual EEG calibration for 5 times a week for 4 weeks
  Arms: RecoveriX with individual EEG calibration
Device: RecoveriX without individual EEG calibration — RecoveriX applied FES according to the brainwave of other subjects regardless of the individual brainwave for 5 times a week for 4 weeks
  Arms: RecoveriX without individual EEG calibration

SUMMARY:
Determination of clinical effects of brain machine interface in chronic stroke patient without wrist extensor strength

DETAILED DESCRIPTION:
The purpose of this study is to compare RecoveriX with individual EEG calibration and without individual EEG calibration to determine the clinical effect of brain machine interface in chronic stroke patient without wrist extensor strength

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Weak wrist extension
* Onset ≥ 6 months
* Fugl-Meyer Assessment score ≥ 19
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* Wrist extensor spasticity above or modified ashworth scale 2
* Severe upper extremity pain that could interfere with rehabilitation therapy
* Neurological disorders other than stroke that can cause motor deficits
* Uncontrolled severe medical conditions.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - upper extremity | 4 weeks after baseline
  Fugl-Meyer Assessment is indicator of the level of impairment of upper extremity, with higher scores indicating lower impairment.
  Total scores range from 0 to 66, each item being scored on a 3-point scale (0, cannot perform; 1, partially performs; and 2, fully performs the task).

SECONDARY OUTCOMES:
Box and block test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Box and block test measures unilateral gross manual dexterity. Higher scores indicate better gross manual dexterity.
Jebsen hand function test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Jebsen hand function test provides a standardized and objective evaluation of fine and gross motor hand function using simulated activities of daily living. Total score is the sum of time taken for each subtest, which are rounded to the nearest second. Shorter times indicate better performance.
9-hole peg test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  9-hole peg test measures finger dexterity in patients with stroke. Scores are based on the time taken to complete the test activity, recorded in seconds.
Medical Research Council (MRC) scale of affected upper extremity | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  The MRC is a standardized set of assessments that measure muscle strength and function.
  The MRC scale of muscle strength uses a score of 0 to 5 to grade the power of a particular muscle group in relation to the movement of a single joint.
Joint position sense | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Joint position sense is tested by holding the most distal joint of a digit by its sides and moving it slightly up or down. First, demonstrate the test with the patient watching so they understand what is wanted then perform the test with their eyes closed.
Sensation of limb movement | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  For the ability to sense a sharp object, the best screening test uses a safety pin or other sharp object to lightly prick the face, torso, and 4 limbs; the patient is asked whether the pinprick feels the same on both sides and whether the sensation is dull or sharp.
active range of motion (AROM) of wrist flexion/extension | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  active range of motion of wrist flexion and extension
Modified Ashworth scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Modified Ashworth scale measures resistance during passive soft-tissue stretching.
  Scores range from 0-4, with 5 choices. A score of 1 indicates no resistance, and 5 indicates rigidity.
Stroke impact scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Stroke impact scale evaluates how stroke has impacted your health and life. Each item is rated in a 5-point Likert scale in terms of the difficulty the patient has experienced in completing each item. Summative scores are generated for each domain, scores range from 0-100.
electroencephalography (EEG) effective connectivity | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  EEG effective connectivity describes the causal influences that neural units exert over another.
Stroke rehabilitation motivation scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Stroke rehabilitation motivation scale includes 28 items applicable to stroke rehabilitation, adapted from the Sports Motivation Scale. The response to each item is measured on a scale of 1 to 5. Higher score indicates higher rehabilitation motivation level for all items, except three reverse evaluation items (items #5, #12, and #23), for which a higher score indicates lower motivation level.
Intrinsic motivation inventory | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  The Intrinsic Motivation Inventory assesses participants' interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice while performing a given activity, thus yielding six subscale scores. A higher score will indicate more of the concept described in the subscale name.
Motor evoked potential | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  action potential elicited by noninvasive stimulation of the motor cortex through the scalp

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea